CLINICAL TRIAL: NCT00266110
Title: Phase II Trial Evaluating the Toxicity and Efficacy of a Multiepitope Dendritic Cell Vaccine Given With Trastuzumab and Vinorelbine Ditartrate for the Treatment of Women With Metastatic Breast Cancer That Express HLA-A0201 and Whose Tumors Overexpress HER-2/NEU
Brief Title: Vaccine Therapy, Trastuzumab, and Vinorelbine in Treating Patients With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0418; P50CA058223 (NIH); R21CA105837 (NIH); KG100307 (Other Grant/Funding Number: Susan G Komen for the Cure)
Record Dates: First submitted 2005-12-13; First posted 2005-12-15 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sargramostim; Trastuzumab; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dendritic Cell Vaccine (Experimental): Therapeutic autologous dendritic cells (Dendritic Cell Vaccine) i.d. injection, 20 x 106 DCs given per treatment Trastuzumab infusion Vinorelbine ditartrate infusion
  Interventions: Biological: sargramostim; Biological: therapeutic autologous dendritic cells; Biological: trastuzumab; Drug: vinorelbine ditartrate

INTERVENTIONS:
Biological: sargramostim — All patients will receive Leukine (GM-CSF) at 250 mcg/m2 starting one day after the administration of chemotherapy x 7 days. Patients with neutrophil counts below 1,000/mm3 on day 8 will continue GM-CSF therapy until the neutrophil count is greater than 1,000/mm3.
  Other Names: Leukine
Biological: therapeutic autologous dendritic cells — patients will receive (10 x 106) peptide-pulsed DCs given by i.d injection into either axilla or the inguinal region with each peptide given into a separate site. The total dose will be 20 x 106 DCs given per treatment.
Biological: trastuzumab — Trastuzumab will be infused in the side-port of a freely flowing IV over 90 minutes and at 6mg/kg if the subject has not previously received Trastuzumab, or if it has been more than 30 days since any prior trastuzumab administration. If the subject has previously received Trastuzumab within 30 days and has no adverse history with the drug, the infusion will be given over 30 minutes. If the subject is currently receiving Trastuzumab, the first study infusion will be given at 4mg/kg over 30 minutes. Subsequently, Trastuzumab will be infused at 4 mg/kg in the side-port of a freely flowing IV over 30 minutes.
  Other Names: Herceptin
Drug: vinorelbine ditartrate — Vinorelbine 25 mg/m2 will be administered IV over six to ten minutes into the side port of a freely flowing IV line.
  Other Names: Navelbine

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells may help the body build an effective immune response to kill tumor cells. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving vaccine therapy together with trastuzumab and vinorelbine may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving vaccine therapy together with trastuzumab and vinorelbine works in treating patients with locally recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of multiepitope autologous dendritic cell vaccine in combination with trastuzumab (Herceptin®) and vinorelbine ditartrate in patients with locally recurrent or metastatic breast cancer whose tumors overexpress human epidermal growth factor receptor 2 (HER2/neu).

Secondary

* Determine if this regimen is effective in generating functional antigen-specific T cells.

OUTLINE:

* Therapeutic autologous dendritic cell (DC) preparation: Patients undergo mobilization of DC and apheresis for production of therapeutic DC. DCs are expanded in vitro for 10-20 days and pulsed with E75 and E90 peptides.
* Treatment: Patients receive vinorelbine ditartrate IV over 6-10 minutes, therapeutic autologous DC intradermally over 2-5 minutes, and trastuzumab (Herceptin®) IV over 30-90 minutes on day 1. Patients receive sargramostim (GM-CSF) subcutaneously on days 2, 4, and 6, or until neutrophil counts recover. Treatment repeats every 14 days for up to 6 courses (or more at the discretion of the investigator) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
PATIENT ELIGIBILITY

4.1 Inclusion Criteria 4.1.1 Histologically proven metastatic breast cancer with measurable or evaluable disease per investigator discretion.

4.1.2 Patients must be 18 years of age or older. Women of child bearing potential must be practicing barrier or oral contraception for the duration of the study, or documented as surgically sterile or one year post-menopausal.

4.1.3 Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (See Appendix A).

4.1.5 Cardiac function by multigated acquisition scan (MUGA) with an ejection fraction (EF) > 45% or an echocardiogram that shows normal left ventricle (LV) function.

4.1.6 Serum Creatinine < 2.0 mg/dl. 4.1.7 Hepatic transaminases (alanine aminotransferase (ALT) and aspartate aminotransferase (AST)) ≤3.0 times the upper limit of normal if no liver metastases or ≤5 times the upper limit of normal if liver metastases are present.

4.1.8 Bilirubin no more than 2 times normal.

4.1.9 Seronegative for HIV.

4.1.10 Negative for Hepatitis B surface antigen.

4.1.11 Signed and dated informed consent.

4.1.12 HLA A0201+ by DNA genotyping.

4.1.13 Absolute neutrophil count greater than 1,500/mm3. Platelet count greater 100,000/mm3 and hemoglobin greater than or equal to 10

4.1.14. 3+ expression of HER-2/neu from original pathology (diagnostic) tumor sample by Immunohistochemistry (IHC) or 2+ expression by IHC with gene amplification by fluorescence in situ hybridization (FISH).

4.1.15. Patients will be eligible even if they have failed treatment for metastatic breast cancer with trastuzumab and a chemotherapy agent other than vinorelbine or if they have progressed within 12 months of receiving adjuvant chemotherapy using trastuzumab and a taxane.

4.2 Exclusion Criteria

4.2.1 Patients with any serious medical, cardiac, or psychiatric condition which, in the opinion of the investigator, would make the patient unsuitable for study participation or would impede probable compliance with the protocol.

4.2.2 Patients with central nervous system metastases must have stable disease for at least 3 months prior to study entry.

4.2.3 Patient is currently taking steroid medications. Systemic steroid treatment is not allowed.

4.2.4 Patients that have failed prior therapy with vinorelbine + trastuzumab will not be eligible for therapy.

4.2.5 Patient has received hormonal or cytotoxic chemotherapy within 14 days of apheresis and within 28-30 days prior to study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2017-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S. Serody, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: web address for Lineberger Comprehensive Cancer Center, University of North Carolina (UNC) — http://www.unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from University of North Carolina (UNC) at Chapel Hill.
Pre-assignment Details: 105 patients were consented for this study, 103 were on-study, and 17 began treatment.
Groups:
- Dendritic Cell Vaccine: Therapeutic autologous dendritic cells (Dendritic Cell Vaccine) i.d. injection, 20 x 106 DCs given per treatment Trastuzumab infusion Vinorelbine ditartrate infusion
  Sargramostim: All patients will receive Leukine (GM-CSF) at 250 mcg/m2 starting one day after the administration of chemotherapy x 7 days. Patients with neutrophil counts below 1,000/mm3 on day 8 will continue GM-CSF therapy until the neutrophil count is greater than 1,000/mm3.
  Therapeutic autologous dendritic cells: patients will receive (10 x 106) peptide-pulsed dendritic cells (DCs) given by i.d injection into either axilla or the inguinal region with each peptide given into a separate site. The total dose will be 20 x 106 DCs given per treatment.
  Trastuzumab: Trastuzumab will be infused in the side-port of a freely flowing IV over 90 minutes and at 6mg/kg if the subject has not previously received Trastuzumab, or if it has been more than 30 days since any prior trastuzumab administration.
Period: Overall Study
Arm/Group | Dendritic Cell Vaccine
Started | 17
Completed | 10
Not Completed | 7

BASELINE CHARACTERISTICS:
Groups:
- Dendritic Cell Vaccine: Therapeutic autologous dendritic cells (Dendritic Cell Vaccine) i.d. injection, 20 x 106 DCs given per treatment Trastuzumab infusion Vinorelbine ditartrate infusion
  sargramostim: All patients will receive Leukine (GM-CSF) at 250 mcg/m2 starting one day after the administration of chemotherapy x 7 days. Patients with neutrophil counts below 1,000/mm3 on day 8 will continue GM-CSF therapy until the neutrophil count is greater than 1,000/mm3.
  therapeutic autologous dendritic cells: patients will receive (10 x 106) peptide-pulsed DCs given by i.d injection into either axilla or the inguinal region with each peptide given into a separate site. The total dose will be 20 x 106 DCs given per treatment.
  trastuzumab: Trastuzumab will be infused in the side-port of a freely flowing IV over 90 minutes and at 6mg/kg if the subject has not previously received Trastuzumab, or if it has been more than 30 days since any prior trastuzumab administration.
Arm/Group | Dendritic Cell Vaccine
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 65.18 [47 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: Response: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 5-6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dendritic Cell Vaccine
Number analyzed (Participants) | 17
Participants | 0

2. Secondary Outcome: Generation of E75/E90 Tetramer-positive CD8+ T Cells
Description: Evaluate the ability of peptide-pulsed dendritic cells plus trastuzumab to induce functional antigen specific T cells. Measured by percentage of intracellular cytokine staining for E75/E90 tetramer-positive CD8+ T cells
Time Frame: 13 weeks
Population: One patient failed to have blood drawn for correlative studies following second vaccine.
Measure: Mean (Full Range); unit: Percentage
Groups:
- Dendritic Cell Vaccine: Experimental: Dendritic Cell Vaccine
  Therapeutic autologous dendritic cells (Dendritic Cell Vaccine) i.d. injection, 20 x 106 DCs given per treatment Trastuzumab infusion Vinorelbine ditartrate infusion
Arm/Group | Dendritic Cell Vaccine
Number analyzed (Participants) | 16
Percentage | 3.63 [.17 to 19.4]

3. Secondary Outcome: Generation of Interferon Gamma Positive CD8+T Cells
Description: Evaluate the ability of peptide-pulsed dendritic cells plus trastuzumab to induce functional antigen specific T cells. Measured by percentage of intracellular cytokine staining for interferon gamma positive CD8+ T cells
Time Frame: 13 weeks
Population: Three subjects had insufficient samples due to early withdraw from study, and one subject was removed from study before the vaccine was administered.
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | Dendritic Cell Vaccine
Number analyzed (Participants) | 13
percentage of cells | 15.99 [0.93 to 36.7]

ADVERSE EVENTS:
Time Frame: Toxicity was assessed for 16 weeks.
Arm/Group | Dendritic Cell Vaccine
All-Cause Mortality (participants affected / at risk) | 15/17
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dendritic Cell Vaccine (N=17)
Nausea (Gastrointestinal disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dendritic Cell Vaccine (N=17)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3
Creatinine (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 5
Hypotension (Vascular disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Abdomen NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 1
Injection site reaction/extravasation changes (General disorders) | 1
Insomnia (Psychiatric disorders) | 1
Leukocytes (total WBC) (Investigations) | 4
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2
Mood alteration - Anxiety (Psychiatric disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 3
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 2
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1
Platelets (Investigations) | 1
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 4
Rigors/chills (General disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1
Taste alteration (dysgeusia) (Nervous system disorders) | 1
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 2
Weight loss (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes